CLINICAL TRIAL: NCT02429414
Title: Prospective Randomized Study on Video Double-Lumen Tube Versus Double-Lumen Tube
Brief Title: Video Double-Lumen Tube Prospective Randomized Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: E.T. View Medical Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-0991; NCI-2015-01551 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Results first posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Other Surgical Procedures
Keywords: Surgical Procedure; Fiberoptic bronchoscopy; FOB; Non-Video Double Lumen Tube; DLT; Video Double Lumen Tube; VDLT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Non-Video Double Lumen Tube (DLT) Group (Experimental): Participants receive a non-video DLT for lung isolation before surgery. Once non-video DLT is in correct place, its final position before surgery checked with a fiberoptic bronchoscopy (FOB).
  Interventions: Device: Non-Video Double Lumen Tube (DLT); Procedure: Fiberoptic Bronchoscopy (FOB)
- Video Double Lumen Tube (VDLT) Group (Experimental): Participants receive a VDLT for lung isolation before surgery. Once VDLT is in correct place, its final position before surgery checked with the camera inside the tube.
  Interventions: Device: Video Double Lumen Tube (VDLT)

INTERVENTIONS:
Device: Non-Video Double Lumen Tube (DLT) — Participant receives non-video double lumen tube (DLT) placement before surgery.
  Other Names: DLT
  Arms: Non-Video Double Lumen Tube (DLT) Group
Procedure: Fiberoptic Bronchoscopy (FOB) — Fiberoptic bronchoscopy (FOB) performed to check placement of non-video DLT.
  Other Names: FOB
  Arms: Non-Video Double Lumen Tube (DLT) Group
Device: Video Double Lumen Tube (VDLT) — Participant receives video double lumen tube (VDLT) placement before surgery.
  Other Names: VDLT
  Arms: Video Double Lumen Tube (VDLT) Group

SUMMARY:
The goal of this clinical research study is to learn how often a fiberoptic bronchoscopy (FOB -- also known as a fiberoptic scope procedure) needs to be used with a video double lumen tube (VDLT) during surgeries that require lung isolation. On this study, you will have one of 2 types of commonly-used breathing tubes used, either a VDLT or a non-video double lumen tube (called a non-video DLT). An FOB may or may not be performed, as described below.

The level of effectiveness of the VDLT and non-video DLT will be compared.

DETAILED DESCRIPTION:
The difference between the 2 types of breathing tubes is that the VDLT has a built-in camera that is designed to allow the doctor to see the airways continuously.

A fiberoptic scope is a thin device that may be placed into the breathing tube in order to check that the tube is in the correct place.

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group. You will have an equal chance of being assigned to either group.

If you are in Group 1, you will receive a non-video DLT for lung isolation before surgery. Once the doctor thinks the non-video DLT is in the correct place, its final position before surgery will be checked with an FOB.

If you are in Group 2, you will receive a VDLT for lung isolation before surgery. Once the doctor thinks the VDLT is in the correct place, its final position before surgery will be checked with the camera inside the tube. However, if the doctor thinks it is needed, an FOB may also be used to confirm that the VDLT is in the correct place.

You will sign a separate consent form that describes the risks of surgery.

Procedures:

Once the doctor thinks the VDLT or non-video DLT is in the correct place and your lung(s) can be isolated, you will have surgery as planned. At the end of surgery, the breathing tube will be removed.

If the breathing tube cannot be placed, you will not have the surgery at that time.

Length of Study:

After the surgery, your study participation will be over.

This is an investigational study. The VDLT and non-video DLT are FDA approved and commercially available. Comparing them is investigational. The study doctor can explain how the study devices are designed to work.

Up to 80 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients need lung isolation for purposed surgery
2. 18 years or older
3. All patients to give written informed consent to participate

Exclusion Criteria:

1. Patient with known tracheobronchial anatomical anomalies
2. Patient requiring emergency operations
3. Patients with known difficult airways
4. Patients where other lung isolation devices may be warranted (tracheostomy, nasal intubation)
5. Patient requiring sizes not available in DLT or VDLT
6. Patients requiring a right sided VDLT or DLT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jagtar S. Heir, DO, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 2015 - July 2016
Pre-assignment Details: 83 participants consented, 3 were not eligible due to (1) withdrew consent, (1) withdrawal by subject, and (1) physician's decision.
Groups:
- Mallinckrodt Double Lumen Tube (DLT): Participants receive a non-video DLT for lung isolation before surgery. Once non-video DLT is in correct place, its final position before surgery checked with a fiberoptic bronchoscopy (FOB). Non-Video Double Lumen Tube (DLT): Participant receives non-video double lumen tube (DLT) placement before surgery. Fiberoptic Bronchoscopy (FOB): Fiberoptic bronchoscopy (FOB) performed to check placement of non-video DLT. Under General Anesthesia, the Double Lumen Tube (DLT) was inserted with conventional laryngoscopy or video laryngoscopy as per the preference of the anesthesiologist. Attending anesthesiologists performed all the intubations.
- Vivasight Video Double Lumen Tube (VDLT): Participants receive a VDLT for lung isolation before surgery. Once VDLT is in correct place, its final position before surgery checked with the camera inside the tube. Video Double Lumen Tube (VDLT): Participant receives video double lumen tube (VDLT) placement before surgery. Under General Anesthesia, the Video Double Lumen Tube (VDLT) was inserted with conventional laryngoscopy or video laryngoscopy as per the preference of the anesthesiologist. Attending anesthesiologists performed all the intubations. Prior to insertion, the VDLT was connected to its accompanying external monitor via a mini universal serial bus port.
Period: Overall Study
Arm/Group | Mallinckrodt Double Lumen Tube (DLT) | Vivasight Video Double Lumen Tube (VDLT)
Started | 42 | 38
Completed | 42 | 37
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mallinckrodt Double Lumen Tube (DLT) | Vivasight Video Double Lumen Tube (VDLT) | Total
Number analyzed (Participants) | 42 | 38 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 23 | 43
  >=65 years | 22 | 15 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 10 | 33
  Male | 19 | 28 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 42 | 38 | 80
American Society of Anesthesiologist (ASA) Status [Count of Participants; unit: Participants] — The ASA (American Society of Anesthesiology) score is a metric to determine if someone is healthy enough to tolerate surgery and anesthesia.
  ASA I A normal healthy patient ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life
  Participants
    ASA I | 1 | 0 | 1
    ASA II | 7 | 11 | 18
    ASA III | 34 | 25 | 59
    ASA IV | 0 | 2 | 2
Mallampati [Count of Participants; unit: Participants] — Class 1-complete visualization of the soft palate, Class II-complete visualization of the uvula, Class III- visualization of only the base of the uvula, and Class IV- soft palate is not visible at all.
  Participants
    Class I | 12 | 5 | 17
    Class II | 24 | 25 | 49
    Class III | 6 | 6 | 12
    Class IV | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fiberoptic Use During Surgeries Requiring Lung Isolation
Description: The rate of FOB use for the VDLT arm and the Double-Lumenendobronchial Tubes (DLT) arm was calculated. The Fisher's exact test or chi-square test was used to evaluate the association between 2 categorical variables. Wilcoxon rank-sum test was used to evaluate the difference in a continuous variable. Rate of fiberoptic use with the Video Double-Lumen Tube (VDLT) during surgeries requiring lung isolation and to compare to the rate of Fiberoptic Bronchoscopy (FOB) use with the conventional DLT.
Time Frame: During surgery (from induction to extubation), an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mallinckrodt Double Lumen Tube (DLT) | Vivasight Video Double Lumen Tube (VDLT)
Number analyzed (Participants) | 42 | 38
Participants | 42 | 5
Statistical Analysis 1: Comparison: Mallinckrodt Double Lumen Tube (DLT) vs Vivasight Video Double Lumen Tube (VDLT); Test type: Superiority; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Quality of View Provided by the VDLT (Embedded Camera) vs. DLT (FOB) Using Grading System
Description: Good is defined as able to visualize all structures and good lung isolation position verified Adequate is defined as able to visualize primary carina, other structures challenging to visualize good lung isolation position verified Poor is defined as unable to recognize anatomy.
Time Frame: During surgery (from induction to extubation), an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mallinckrodt Double Lumen Tube (DLT) | Vivasight Video Double Lumen Tube (VDLT)
Number analyzed (Participants) | 42 | 38
Participants
  Good view | 42 | 33
  Adequate view | 0 | 5
  Poor | 0 | 0
Statistical Analysis 1: Comparison: Mallinckrodt Double Lumen Tube (DLT) vs Vivasight Video Double Lumen Tube (VDLT); Test type: Superiority; p = 0.0209, t-test, 2 sided

3. Secondary Outcome: Number of Participants in Which Anesthesiologist Was Able to Forewarn/ Anticipate Dislodging of Endobronchial Cuff
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Mallinckrodt Double Lumen Tube (DLT) | Vivasight Video Double Lumen Tube (VDLT)
Number analyzed (Participants) | 42 | 38
Participants | 2 | 7
Statistical Analysis 1: Comparison: Mallinckrodt Double Lumen Tube (DLT) vs Vivasight Video Double Lumen Tube (VDLT); Test type: Superiority; p = 0.078, t-test, 2 sided

4. Secondary Outcome: Dislodgement During Positioning and Surgery
Time Frame: During positioning, up to 30 minutes and during surgery (from induction to extubation), up to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mallinckrodt Double Lumen Tube (DLT) | Vivasight Video Double Lumen Tube (VDLT)
Number analyzed (Participants) | 14 | 13
Participants
  Positioning | 9 | 8
  Surgery | 3 | 5

ADVERSE EVENTS:
Time Frame: During surgery (from induction to extubation)
Arm/Group | Mallinckrodt Double Lumen Tube (DLT) | Vivasight Video Double Lumen Tube (VDLT)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/38
Other Adverse Events (participants affected / at risk) | 0/42 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT02429414/Prot_SAP_000.pdf